CLINICAL TRIAL: NCT05180864
Title: Omentum Preservation Versus Complete Omentectomy in Gastrectomy for Gastric Cancer
Acronym: OMEGA-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC (Other)
Responsible Party: Principal Investigator, Suzanne S. Gisbertz, Principal Investigator, Amsterdam UMC, location VUmc
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VUmc_2021-5603
Record Dates: First submitted 2021-06-03; First posted 2022-01-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stomach Neoplasm
Keywords: Gastrectomy; Omentectomy; Survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complete omentectomy (Active Comparator): Gastrectomy with complete omentectomy
  Interventions: Procedure: Gastrectomy
- Omentum presevation (Experimental): Gastrectomy with preservation of the omentum distal to the gastroepiploic vessels
  Interventions: Procedure: Gastrectomy

INTERVENTIONS:
Procedure: Gastrectomy — Open or minimally invasive (sub)total gastrectomy

SUMMARY:
Curative therapy for gastric cancer usually consists of perioperative chemotherapy and a radical (R0) gastrectomy. A radical resection includes a modified D2 lymphadenectomy, and, generally, a complete omentectomy, to ensure the removal of omental metastatic lymph nodes and tumor deposits.

The omentum has some essential functions within the peritoneal cavity. The omentum functions as regulator of regional immune responses to prevent infections and, additionally, it prevents adhesions that can lead to small bowel obstruction. Omentectomy is associated with increased incidence of early and late postoperative complications such as abdominal abscess, ileus, and wound infections in various types of surgery.

There is little evidence regarding survival benefit of routine complete omentectomy during gastrectomy. The investigators hypothesize that omitting a complete omentectomy (and instead preserve the greater omentum distal of the gastroepiploic arcade) during gastrectomy for cancer does not negatively impact survival.

OMEGA is a randomized controlled, open, parallel, non-inferiority, multicenter trial. Adult patients (>18 years) with primary resectable gastric cancer, clinical stage T2-4a N0-3 M0 or cT1N+ scheduled for open or minimally invasive (sub)total gastrectomy are included. The primary study objective is to investigate whether omentum preservation in gastrectomy for cancer is non-inferior to complete omentectomy in terms of three-year overall survival.

DETAILED DESCRIPTION:
Primary objective:

The primary study objective is evaluate whether preservation of the omentum distal to the gastroepiploic vessels in gastrectomy for cancer is non-inferior to complete omentectomy in terms of three-year overall survival.

Secondary objectives:

Comparing the two study arms with regard to:

* Operating time
* Intraoperative blood loss
* Intraoperative complications
* Postoperative complications, defined according to the Clavien-Dindo classification25 and comprehensive complication index (CCI)
* Distribution of lymph node metastases
* R0-resection rate
* Rate of malignant cells in cytology
* Molecular sub classification of gastric cancer
* ICG fluorescent enhancement of omentum in omentum preservation group (in centers that have ICG fluorescence available)
* Protocol compliance to allocated treatment
* Hospital stay, defined as time interval between date of surgery and date of hospital discharge
* Readmission rate within 30-days after surgery
* Reintervention rate within 30-days after surgery
* Reoperation rate within three years after surgery
* Quality of life at baseline, 3, 6, 9, 12 and 24 months, the following questionnaires will be used: EQ-5D-5L, QLQ-C30, QLQ-OG25, CIPN, Happiness, HADS and work productivity
* 3- & 5-year disease-free survival, defined as the period of time from operation to locoregional recurrence, peritoneal recurrence, distant metastases, second gastric cancer or death from any cause. Patients alive and free of all these events will be censored at the last follow-up.
* 5-year overall survival, defined as the period of time from operation to death from any cause. Patients alive and free of all these events will be censored at the last follow-up.
* Cost-effectiveness

Study design:

OMEGA is a randomized controlled, open, parallel, non-inferiority, multicenter trial. Eligible patients have to be operable (ASA <4) with resectable (≦cT4aN3bM0) gastric cancer. Patients will be randomized in a 1:1 ratio between radical (sub)total gastrectomy with omentum preservation or complete omentectomy. Patients will be stratified according to center, neoadjuvant therapy and type of surgery (total or subtotal gastrectomy). The primary endpoint is overall survival at three-years after the operation. In total, 654 patients will be randomized.

Sample size:

The primary endpoint is three-year overall survival. According to survival numbers from the Dutch Cancer Registry (NKR), three-year overall survival after gastrectomy is approximately 50% in the Netherlands. Under the common assumption of exponential survival times, a hazard ratio of 0.862 under the alternative hypothesis, at least 50% and 45% expected events (i.e., death) in the control arm and experimental arm, respectively, at the minimum follow-up of three years, 298 events are needed in total to achieve 80% power at a one-sided significance level of 5% with a non-inferiority hazard ratio of 1.15 (PASS 15 Power Analysis and Sample Size Software (2017). NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass), resulting in 314 patients per study arm. Dropouts will be rare (mostly due to loss to follow-up, which is quite rare in cancer patients), with proportion dropping out expected to be at most 5%. After correction for drop-out we plan to include 327 patients in each of the two arms (654 in total).

Statistical analysis:

Primary endpoint: Descriptive statistics will be calculated to summarize patients' groups included in each of trial arms.

Mean and standard deviation will be presented for normally distributed continuous variables. Median plus interquartile-range (IQR) will be presented continuous variables that are skewed and for ordinal variables. Dichotomous and nominal data will be summarized by means of frequencies and percentages.

Non-inferiority of the experimental treatment in terms of overall survival will be tested using Cox-regression. Non-inferiority will be concluded if the upper limit of the 90% confidence interval falls below the non-inferiority hazard ratio of 1.15, corresponding to a one-sided non-inferiority test at significance level of 5%. Survival will be presented graphically using Kaplan-Meier curves. All analyses will be according to the intention to treat principle. A per protocol analysis will also be performed. The experimental treatment will be declared non-inferior if non-inferiority is shown in both the intention to treat and the per protocol analysis.

Secondary endpoint: as independent samples t-test for normally-distributed continuous outcomes, Mann-Whitney tests for continuous outcomes that are not normally distributed or ordinal outcomes. Categorical outcomes will be compared using chi-square test or Fisher's exact test in case of low (expected) cell counts. Repeatedly measured outcomes will be compared between arms using linear mixed models. Secondary time-to-event outcomes will be compared the using log-rank test. Secondary endpoints will be tested at a two-sided significance level of 5%. Effect sizes suitable for the type of outcome measure will be provided (mean differences, ratio of geometric means, relative risks, hazard ratios) together with their 95% confidence interval.

Subgroup analysis for the effect of experimental treatment on overall survival will be performed for the follow subgroups: patient characteristics (age, male/female), diffuse/intestinal type gastric tumor, subtotal/total gastrectomy, and minimally invasive/open gastrectomy. Effect modification will use Cox regression with the subgroup variable, the arm and their two-way interaction. Additionally, stratified analyses will be performed where HR is calculated separately in each of the subgroups.

Quality of life data will be graphically represented across all time points and analyzed according to the manuals and will presented as domain and summarized scores. Questionnaire outcome comparisons will be analyzed using linear mixed models.

ELIGIBILITY:
Inclusion criteria

* Primary resectable gastric adenocarcinoma, clinical stage T1-4aN0-3M0
* ASA 1-3 (able to undergo surgery)
* Scheduled for open or minimally invasive (sub)total gastrectomy with modified D2-lymphadenectomy, with or without perioperative chemotherapy
* Age above 18
* Able to complete questionnaires in Dutch, English or Italian
* Written informed consent
* Esophageal invasion < 2 cm defined from the upper margin of the gastric rugae as determined by endoscopy

Exclusion Criteria:

* Gastric cancer clinically staged as T1N0
* Locally advanced gastric cancer requiring multi-visceral resection
* Pregnancy
* Previous malignancy (excluding non-melanoma skin cancer, pancreatic neuroendocrine tumor (pNET) <2cm, and gastrointestinal stromal tumor (GIST) <2cm), unless no evidence of disease and diagnosed more than three years before diagnosis of gastric cancer, or with a life expectancy of more than five years from date of inclusion
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator
* Previous gastric or omental surgery, with the exclusion of a gastric perforation Indication for thoracotomy/thoracoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years after surgery
  Overall survival is defined as the period of time from operation to death from any cause. Patients alive and free of all these events will be censored at the last follow-up

SECONDARY OUTCOMES:
5-year overall survival | 5 years after surgery
  Defined as the period of time from operation to death from any cause. Patients alive and free of all these events will be censored at the last follow-up
Intraoperative blood loss | Intraoperative
  The volume of blood loss in milliliters during surgery
Postoperative complications | Within 30-days after surgery
  Defined according to the Clavien-Dindo classification and comprehensive complication index (CCI)
Distribution of lymph node metastases | Pathology report 1/2 weeks after surgery
  The distribution of lymph node metastases in gastric cancer
R0-resection rate | Pathology report 1/2 weeks after surgery
  R0-resection rate of the distal and proximal margin, according to the College of American Pathologists
Rate of malignant cells in cytology | Pathology report 1/2 weeks after surgery
  The proportion of patients with malignant cells in peritoneal lavage cytology
Molecular sub classification of gastric cancer | Pathology report 1/2 weeks after surgery
  DNA methylation arrays will be used to classify the gastric tumor into molecular subtypes
Protocol compliance to allocated treatment | Up to 5 years
  The proportion of patients who change from treatment arm
Hospital stay | Up to 5 year
  Defined as time interval between date of surgery and date of hospital discharge
Readmission rate | Within 30-days after surgery
  Rate of readmission
Reintervention rate | Within 30-days after surgery
  Rate of reintervention
Reoperation rate | Within 3 years after surgery
  Rate of reoperation
Quality of life assessment | At baseline, 3, 6, 9, 12 and 24 months
  Quality of life is assessed using the EuroQol-5 Dimension (EQ-5D-5L) descriptive system.
3- & 5-year disease-free survival | After 3 years and 5 years post-operative
  Defined as the period of time from operation to locoregional recurrence, peritoneal recurrence, distant metastases, second gastric cancer or death from any cause. Patients alive and free of all these events will be censored at the last follow-up
Operative time | Intraoperative
  The surgical procedure duration in minutes, defined as time from first incision to last wound closure.
Cost-effectiveness | Up to 3 years post-operative
  Cost-effectiveness will be calculated by comparing the direct medical cost related to both strategies. The cost-effectiveness is compared by assessing cost per QALY.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne S. Gisberts, MD, PhD, Study Chair — Amsterdam UMC; Wietse J. Eshuis, MD, PhD, Principal Investigator — Amsterdam UMC; Mark I. van Berge Henegouwen, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (16):
- University Medical Center of the Johannes Gutenberg University, Mainz, Germany
- Azienda Ospedaliera Universitaria, Siena, Italy
- Netherlands (13):
  - Amsterdam UMC, Amsterdam, North Holland
  - Ziekenhuis Groep Twente, Almelo
  - Antoni van Leeuwenhoek, Amsterdam
  - Gelre ziekenhuis, Apeldoorn
  - Rijnstate ziekenhuis, Arnhem
  - Catharina Ziekenhuis, Eindhoven
  - Universitait Medisch Centrum Groningen, Groningen
  - Zuyderland ziekenhuis, Heerlen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Medisch Centrum, Rotterdam
  - Elisabeth Tweesteden ziekenhuis, Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht
- Oxford University Hospitals, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keywani K, Eshuis WJ, Borgstein ABJ, van Det MJ, van Duijvendijk P, van Etten B, Grimminger PP, Heisterkamp J, Lagarde SM, Luyer MDP, Markar SR, Meijer SL, Pierie JPEN, Roviello F, Ruurda JP, van Sandick JW, Sosef M, Witteman BPL, de Steur WO, Lissenberg-Witte BI, van Berge Henegouwen MI, Gisbertz SS. Omentum preservation versus complete omentectomy in gastrectomy for gastric cancer (OMEGA trial): study protocol for a randomized controlled trial. Trials. 2024 Sep 4;25(1):588. doi: 10.1186/s13063-024-08396-z. PMID 39232781